CLINICAL TRIAL: NCT04222413
Title: First-in-Human Phase I Trial to Investigate the Safety, Tolerability, Pharmacokinetics, Biological and Clinical Activity of Metarrestin (ML-246) in Subjects With Metastatic Solid Tumors
Brief Title: Metarrestin (ML-246) in Subjects With Metastatic Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 200023; 20-C-0023
Record Dates: First submitted 2020-01-07; First posted 2020-01-10 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-09-30

CONDITIONS: Advanced Solid Tumors; Metastatic Pancreatic Cancer; Pediatric Solid Tumor; Advanced Breast Cancer; Malignant Peripheral Nerve Sheath Tumor; Colorectal Neoplasms
Keywords: First-In-Class Investigational Agent; Peri-Nucleolar Compartment (PNC); effective therapies against metastasis; Oral Administration; Maximum Recommended Starting Dose
MeSH Terms: conditions — Pancreatic Neoplasms; Neurofibrosarcoma; Colorectal Neoplasms | interventions — metarrestin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- 1/Arm 1 (Experimental): Escalating/de-escalation doses of metarrestin
  Interventions: Drug: Metarrestin
- 2/Arm 2 (Experimental): MTD of metarrestin
  Interventions: Drug: Metarrestin

INTERVENTIONS:
Drug: Metarrestin — Phase IA: Loading dose on Day 1 of Cycle 1 for Dose Levels 1-7. Loading dose on Days 1 and 3 of Cycle 1 for Dose Levels 8-11. After the loading dose on Day 1 or Days 1 and 3 of Cycle 1, continue on Mondays-Wednesdays-Fridays of every following cycle. Phase IB: PO according to the dose and schedule estimated during Phase IA

SUMMARY:
Background:

Metastasis is the spread of cancer from one organ to a nonadjacent organ. It causes 90% of cancer deaths. No treatment specifically prevents or reduces metastasis. Researchers hope a new drug can help. It stops cancer cells from growing and spreading further and possibly shrink cancer lesions in distant organs.

Objective:

To find a safe dose of metarrestin and to see if this dose shrinks tumors.

Eligibility:

Adults age 18 and older with pancreatic cancer, breast cancer, or a solid tumor that has not been cured by standard therapies. Also, children age 12-17 with a solid tumor (other than a muscle tumor) with no standard therapy options.

Design:

Participants will be screened with:

* blood tests
* physical exam
* documentation of disease confirmation or tumor biopsy
* electrocardiogram to evaluate the heart
* review of their medicines and their ability to do their normal activities

Participants will take metarrestin by mouth until they cannot tolerate it or stop to benefit from it. They will keep a medicine diary.

Participants will visit the Clinical Center. During the first month there are two brief hospital stays required with visits weekly or every other week thereafter. They will repeat some of the screening tests. They will fill out questionnaires. They will have tests of their cognitive function. They will have an electroencephalogram to record brain activity. They will have a computed tomography (CT) scan or magnetic resonance imaging (MRI). A CT is a series of X-rays of the body. An MRI uses magnets and radio waves to take pictures of the body.

Adult participants may have tumor biopsies.

Participants will have a follow-up visit 30 days after treatment ends. Then they will have follow-up phone calls or emails every 6 months for the rest of their life or until the study ends.

DETAILED DESCRIPTION:
Background:

Metarrestin is a first-in-class investigational agent targeting the peri-nucleolar compartment (PNC), a marker of genome organization associated with metastasis.

Preclinical studies have shown that metarrestin effectively suppresses metastasis and extends overall survival in different cancer models.

Multi-species allometric scaling and good laboratory practice (GLP) toxicology and toxicokinetic studies indicate that metarrestin administered at a calculated safe maximum recommended starting dose (MRSD) to human subjects is predicted to afford intratumoral exposure levels within the therapeutic range observed preclinically.

Objectives:

Phase IA: To determine the maximum tolerated dose (MTD) of metarrestin.

Phase IB: To determine the Objective Response Rate (ORR) according to Evaluation Criteria (RECIST 1.1) in patients treated with metarrestin at the MTD.

Eligibility:

Adult subjects with any advanced solid tumors (Cohort IA), or pancreatic, colorectal, or breast tumors (Cohort IB1).

OR

Pediatric subjects age 12 and older with solid tumors other than rhabdomyosarcoma (RMS) including embryonal, alveolar, spindle cell/sclerosing, and pleomorphic subtypes of RMS (Cohort IB2).

Patients must have progressed on prior standard chemotherapeutic therapy.

Design:

This is first-in-human Phase I trial to investigate the safety and clinical activity of metarrestin in subjects with metastatic solid tumors.

During Phase IA MTD of metarrestin will be estimated in adult patients with solid tumors.

During Phase IB adult patients with breast, colorectal, or pancreatic cancer, and pediatric patients with solid organ cancer will be treated at dose level of estimated MTD.

Patients will receive treatment in cycles consisting of 28 (+7/- 2) days.

Metarrestin will be administered PO until progression or unacceptable toxicity.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Adult (>= 18 years) subjects with:

  * histologically or cytologically confirmed solid tumors (Phase IA).

OR

--histologically or cytologically confirmed pancreatic, colorectal, or breast cancer (Phase IB)

OR

* Pediatric (>=12 and < 18 years) subjects with histologically or cytologically confirmed solid tumors other than rhabdomyosarcoma (RMS) including embryonal, alveolar, spindle cell/sclerosing and pleomorphic subtypes of RMS (Phase IB).
* Subjects must have disease that:

  * is not amenable to potentially curative resection,
  * spread at least to one other organ system other than primary tumor or recurred after removal of primary tumor
  * has site measurable per RECIST 1.1
  * progressed on or after at least one line of standard systemic chemotherapy (Phase IA and IB1)
  * have no standard therapy option available (Phase IB2)
* Patients must have recovered from any acute toxicity related to prior therapy or surgery or disease to a grade 1 or less.
* Performance status

  --Karnofsky >= 70% (for patients >= 16 years old), Lansky >= 70% (for patients <16 years old)
* Adequate hematological function defined by:

  * absolute neutrophil count (ANC) >= 1.0 x 10(9)/L,
  * transfusion-independent platelet count >= 100 x 10(9)/L,
  * Hgb >= 9 g/ dL (patients who have received <= 2 PRBC transfusions within 48 hours are eligible)
* Adequate coagulation as defined by:

  --INR<1.5 (or < 3.0 if subjects are currently taking anticoagulated medications) Note: increase of the upper limit of INR is restricted only to subjects who are receiving anticoagulation for medical reasons (DVT/PE prophylaxis, treatment for a thromboembolic event) and have increased INR because of these medications. Patients who have an elevated INR due to compromised liver function or any other medical conditions remain excluded
* Adequate hepatic function defined by:

  * a total bilirubin level <= 1.5 x ULN, (total bilirubin <= 2.0 x ULN in case of prior diagnosis of Gilbert syndrome)
  * an AST level <= 3xULN
  * an ALT level <= 3 xULN
* Adequate renal function defined by:

  * Creatinine OR Measured or calculated creatinine clearance (CrCl) (eGFR may also be used in place of CrCl)

    ---< 1.5x institution upper limit of normal OR

    --->= 45 mL/min/1.73 m^2 for participant with creatinine levels >= 1.5 X institutional ULN
  * Creatinine clearance (CrCl) or eGFR should be calculated per institutional standard.
* The effects of the study treatment on the developing human fetus are unknown; thus, individuals of childbearing potential and individuals who can father children must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior

to study entry, for the duration of study therapy and up to 120 days after the last dose of the study drug.

* Nursing participants must be willing to discontinue nursing at the time of the study treatment initiation.
* Weight >= 35 kg.
* Ability of subject or parent/guardian to understand and the willingness to sign a written informed consent document.
* Subjects must have lesion(s) accessible for biopsy (other than used for measurement of disease) and be willing to undergo mandatory study biopsies (Cohort IB1 only).
* Ability to swallow oral capsules.

EXCLUSION CRITERIA:

* Anticancer treatment within designated period before treatment initiation including:

  * minor surgical procedure (such as biliary stenting) within 14 days. Note: if liver function tests after biliary stenting or renal function tests after ureteral stenting return to normal, within 5 days after biliary or ureteral stenting;
  * major surgical procedure or curative radiation treatment within 28 days;
  * palliative radiation treatment within 14 days;
  * chemotherapy or experimental drug treatment with published half-life known to be 72 hours or less within 14 days;
  * experimental drug treatment with unpublished or half-life greater than 72 hours within 28 days;
  * chemotherapy regimen containing an alkylating antineoplastic agent (cyclophosphamide, chlorambucil, melphalan, or ifosfamide), alkylating-like (platinumbased chemotherapeutic drugs, platinum analogues), and non-classical alkylating agent (dacarbazine, temozolomide) within 28 days.
* Patients receiving any medications or substances that are moderate and strong inhibitors or inducers of CYP3A4 and are not able to safely stop these medications are excluded from this study; patients must stop strong CYP3A4 inhibiting/inducing medications within 5 published half-lives and moderate within 3 published half-lives prior to the treatment initiation.

Note: dihydropyridine calcium - channel blockers are permitted for management of underling disease

* Subjects with cardiomyopathy diagnosed within 6 months prior to treatment initiation including but not limited to the following:

  * hypertrophic cardiomyopathy
  * arrhythmogenic right ventricular cardiomyopathy
  * abnormal ejection fraction (echocardiogram [ECHO]) <= 53% (if a range is given then the upper value of the range will be used)
  * previous moderate or severe impairment of left ventricular systolic function (LVEF <45%)
  * severe valvular heart disease
  * atrial fibrillation with a ventricular rate >100 bpm on EKG at rest
  * Fridericia's corrected QT interval (QTcF) >= 480 msec (adults) or >= 460 msec (pediatric subjects, aged 12 to <18 years) or other factors that increase the risk of QT prolongation or arrhythmic events (e.g., heart failure, hypokalemia, family history of long QT interval syndrome.
* HIV, HCV, HBV positive patients on antiviral drugs are excluded due to the absence of previous experience with concurrent use of antiviral medications and the investigational drug product to be evaluated in the current study and possible for adverse pharmacokinetic and/or pharmacodynamic interactions.
* Previous malignant disease (other than the target malignancy to be investigated in this trial) within the last 3 years. Note: subjects with a history of cervical carcinoma in situ, superficial or non-invasive bladder cancer, or basal cell or squamous cell carcinoma in situ previously treated with curative intent are NOT excluded.
* Rapidly progressive disease which, in the opinion of the Investigator, may predispose to inability to tolerate treatment or trial procedures.
* Subjects with central nervous system (CNS) metastases or CNS disorders known to increase possible neurotoxicity of metarrestin in case of compromised blood-brain barrier (e.g. recent stroke (<3 months of treatment initiation), infectious causes).
* Significant acute or chronic infections including tuberculosis with presence of clinical symptoms or physical findings.
* Patients with a history of any seizures or increased risk of seizures on screening EEGs defined by 1) interictal epileptiform discharges, 2) temporal intermittent rhythmic delta activity (TIRDA), or 3) electrographic or clinical seizures on EEG.
* Clinically relevant diseases (for example, inflammatory bowel disease) and / or uncontrolled medical conditions, which, in the opinion of the Investigator, might impair the subject's tolerance or ability to participate in the trial.
* Patients with previous gastric bypass, patients receiving nutrition via feeding tubes or parenterally, or patients with malabsorptive conditions (damage to the intestine from infection, inflammation, trauma, or surgery, celiac disease, Crohn's disease, chronic pancreatitis, or cystic fibrosis resulting malabsorption). Patients with refractory nausea and vomiting. Note: patients with gastric banding are allowed.
* Pregnant individuals.

Ages: 12 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 116 (Estimated)
Dates: Start 2020-10-27 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
To identify the maximum tolerated dose (MTD) of metarrestin in subjects with metastatic solid tumors | 28 days
  MTD of metarrestin
To determine the Objective Response Rate (ORR) according to Evaluation Criteria (RECIST 1.1) in patients treated with metarrestin at the MTD | every 2 months
  Fraction of objective responses determined and reported as the ORR

SECONDARY OUTCOMES:
To determine the Objective Response Rate (ORR) according to Evaluation Criteria (RECIST 1.1) in patients treated with metarrestin at the MTD in Cohort IB1 | every 2 months
  The ORR rate will be determined by dividing the number of patients with an objective response by the number of evaluable patients who are treated at the MTD for cohort Phase IB1
To determine plasma PK levels of metarrestin in humans | 28 days
  The pharmacokinetic (PK) profile of metarrestin will be derived from single dose and multiple dose PK measures for each dose level collecting the standard pharmacokinetic parameters
To assess progression-free survival (PFS) according to RECIST 1.1 | at progression
  Median amount of time subject survives without disease progression after treatment
To determine duration of overall response (DOR) rate according to Response Evaluation Criteria (RECIST 1.1) in subjects with metastatic solid tumors | at progression
  Kaplan-Meier curves beginning at the date of response will be used and will be determined in all responding patients treated on the Phase IB expansion cohorts
To determine tolerability of the adult recommended dose in children >= 12 year of age (Cohort IB2) | 28 days after treatment discontinuation
  The fraction of patients who can tolerate the dose
To assess safety and tolerability of metarrestin (Cohort IB1) | 28 days after treatment discontinuation
  All treatment-related AEs will be captured, and for each grade, the number and type of AE per dose level will be descriptively described in Cohort 1B1
To assess safety and tolerability of metarrestin in subjects with metastatic solid tumors | 28 days after treatment discontinuation
  All treatment-related AEs will be captured, and for each grade, the number and type of AE per dose level will be descriptively described

CONTACTS AND LOCATIONS:
Overall Officials: Udo Rudloff, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - University of Kansas, Fairway, Kansas
  - National Institutes of Health Clinical Center, Bethesda, Maryland

IPD SHARING:
Plan to Share IPD: Yes
All IPD recorded in the medical record will be shared with intramural investigators upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Clinical data available during the study and indefinitely.
Access Criteria: Clinical data will be made available via subscription to BTRIS and with the permission of the study PI.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?A_2020-C-0023.html